CLINICAL TRIAL: NCT06240364
Title: Effects of AffronEye®/ Crocuvis+® on Dry Eye Syndrome
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alicante (Other)
Collaborators: Pharmactive Biotech Products S.L.U (Industry)
Responsible Party: Principal Investigator, Maria del Mar Seguí Crespo, Senior Lecturer, PhD, University of Alicante
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: PHARMACTIVE1-24I
Record Dates: First submitted 2024-01-22; First posted 2024-02-05 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Dry Eye Syndrome
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Saffron extract (Crocus sativus) (Experimental): Daily intake of one tablet for 84 days.
  Interventions: Dietary Supplement: Saffron extract (Crocus sativus)
- Placebo (Placebo Comparator): Daily intake of one tablet for 84 days. This tablet is organoleptically indistinguishable from the experimental tablet.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Saffron extract (Crocus sativus) — Daily intake of one tablet for 84 days.
  Arms: Saffron extract (Crocus sativus)
Dietary Supplement: Placebo — Daily intake of one tablet for 84 days.
  Arms: Placebo

SUMMARY:
Previous research has demonstrated the effectiveness of AFFRONEYE® / CROCUVIS+® dietary supplement, based on saffron extract, in the proper functioning of visual health, for example, against the development of glaucoma. The main objective of this study is to compare the results of clinical tests that evaluate signs and symptoms for the diagnosis of dry eye, between two groups (some that take the dietary supplement and others a placebo), in a sample of university workers and students who suffer from dry eye.

ELIGIBILITY:
Inclusion Criteria:

* Have dry eye according to the diagnostic criteria established by the Tear Film and Ocular Surface Society (TFOS) Dry Eye Workshop (DEWS).

Exclusion Criteria:

* Pathology of the anterior ocular surface under treatment (such as conjunctivitis, keratitis, among others).
* Take any type of dietary supplements, with or without botanical components in the last month.
* Pregnancy or breastfeeding (also excludes recent pregnancy within the last 3 months) and women planning to become pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2025-10-10 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline dry eye symptoms at 28, 56 and 84 days | 0 (baseline), 28, 56 and 84 days
  Measured with Ocular Surface Disease Index (OSDI, adapted version to spanish). It consists of 12 items that assess symptoms, functional limitations, and environmental factors related to dry eye. The score ranges from 0 to 100 (worst). Each item is evaluated on a 4-point Likert scale (from 0 to 4). The final score is obtained from (the sum of scores for all questions answered x 25) and divide to total number of questions answered (do not included questions answered N/A); dry eye symptoms are considered from ≥ 13 points.
Changes with respect to baseline NIBUT at 28, 56 and 84 days | 0 (baseline), 28, 56 and 84 days
  Non-Invasive tear BreakUp Time (NIBUT). It is measured with the Keratograph 5M topographer. It is used to assess tear film stability. It is a non-invasive method to observe and detect the tear film break-up time (measured in seconds). In this case, fluorescein staining can be dispensed with, thus eliminating any influence it may have on the tear film and the results. The region and time course of tear film rupture are automatically measured without user intervention.
  The software analyses the Placido projecting rings on the tear film and automatically detects any distortion or discontinuity in the reflected annular pattern. The results are recorded with respect to time and space, and translated into a colour-coded map.
  A positive finding has been reported to be a value <10 s.
Changes with respect to baseline TMH at 28, 56 and 84 days | 0 (baseline), 28, 56 and 84 days
  Tear Meniscus Height (TMH). It is measured with the Keratograph 5M topographer. It assesses the height of the lacrimal meniscus (measured in millimetres). Firstly, it provides information on the secretory capacity of the main lacrimal gland and secondly, it may indicate a high evaporation rate, which may, for example, be due to an insufficient lipid layer.
  It is measured with a ruler from the point of the lower lid margin (below the centre of the pupil) to the upper edge of the lacrimal meniscus.
  A positive finding has been reported to be a value <0.2 mm.
Changes with respect to baseline ocular surface stainings at 28, 56 and 84 days | 0 (baseline), 28, 56 and 84 days
  Ocular surface stains are used to assess epithelial damage to the cornea, conjunctiva, and lid margin.
  To assess corneal epithelial damage, a fluorescein strip is wet with saline, and a drop is instilled inside the lower temporal lid. Optimal viewing is 1-3 minutes after instillation. A positive result is >5 corneal spots.
  To assess conjunctival and lid margin damage, a lissamine green strip is wet with saline, and a drop is instilled inside the lower temporal lid. The observation should occur between 1 and 4 min postinstillation.
  To assess conjunctival damage, a positive score is > 9 conjunctival spots. To assess lid margin damage, ≥2 mm in length and/or ≥25% sagittal width is a positive score.
Changes with respect to baseline lipid layer of the tear film at 28, 56 and 84 days | 0 (baseline), 28, 56 and 84 days
  The thickness of the lipid layer is not uniform throughout its structure and is examined by observing an interferential phenomenon with Keratograph 5M topographer.
  The ideal pattern is yellow to blue color at around 80-100nm. If excessively colored patterns are observed, this refers to a greater lipid film thickness >100nm. If, on the other hand, the pattern is gray-white, it indicates a thin or absent lipid layer, causing greater evaporation.
Changes with respect to baseline MGD at 28, 56 and 84 days | 0 (baseline), 28, 56 and 84 days
  Meibomian Gland Dysfunction (MGD). The morphological changes of these glands are evaluated using the Keratograph 5M topographer using integrated infrared diodes that allow illumination of the everted eyelids.
  The Meibomian glands are located in the tarsal conjunctiva of the upper and lower eyelids and have the function of producing an oily substance (meibum), which forms the lipid layer of the tear film, protecting it against evaporation of its aqueous phase.
  The number of meibomian glands should be evaluated in the photographs taken; the larger the area without glands, the greater the DGM.
Changes from baseline osmolarity at 28, 56 and 84 days | 0 (baseline), 28, 56 and 84 days
  Measured with the Tearlab osmometer. A positive result is considered to be ≥308 mOsm/L in either eye or an interocular difference >8 mOsm/L.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alicante, San Vicent del Raspeig, Alicante, Spain

IPD SHARING:
Plan to Share IPD: No